CLINICAL TRIAL: NCT06364618
Title: Use of Continuous Biomonitoring for Detection of Infectious Complications in Kidney Transplant Recipients
Brief Title: Use of Wearables to Detect Infections in Kidney Transplant Recipients
Acronym: RENALERT
Status: Not yet recruiting | Type: Observational
Sponsor: Institute for Clinical and Experimental Medicine (Other Government)
Responsible Party: Principal Investigator, Prof. Ondřej Viklický, M.D., Ph.D., Head of Transplantation Center, Principal Investigator, Institute for Clinical and Experimental Medicine
Other Study IDs: G-24-07
Record Dates: First submitted 2024-04-03; First posted 2024-04-15 (Actual); Last update posted 2024-04-15 (Actual); Status verified 2024-04

CONDITIONS: Kidney Transplant Infection
Keywords: biometric data; continuous monitoring; machine learning; early alert system; infection; kidney transplantation
MeSH Terms: conditions — Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — plasma, serum at enrollment and then ad hoc at infection event
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to develop a machine learning algorithm for early detection of infections in kidney transplant recipients using data recorded by wearable digital health technologies.

The main questions it aims to answer are:

1. What are the biometric data pattern changes in impending infections?
2. What accuracy the machine learning algorithm can achieve?

Participants will be given/use their own wearable device that will record biometric data. Any infection event will be recorded and an algorithm will be trained to recognize changes in biometric data preceding symptomatic infection.

ELIGIBILITY:
Inclusion Criteria:

* kidney transplant recipient
* age 18 years or more
* kidney allograft function (eGFR based on CKD-EPI more than 15ml/min/1.73m2)

Exclusion Criteria:

* recipient of another transplanted organ
* terminal failure of another organ (heart, liver, lung)
* diabetes mellitus type 1
* pregnant or breastfeeding woman
* refusal to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Kidney transplant recipients followed at the Institute for Clinical and Experimental Medicine.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Accuracy of the algorithm at detecting infections at presymptomatic stage | The primary endpoint will be assessed periodically throughout the study, up to 24 months.
  Accuracy, sensitivity, specificity, negative and positive predictive value of the machine learning algorithm at detecting infections in presymptomatic stage in kidney transplant recipients.

OTHER OUTCOMES:
Rate of in-patient admissions | Periodically throughout the study, up to 24 months.
  Any hospital admission for infection treatment is considered an event of this outcome
Incidence of decrease/increase of Quality of Life | Periodically throughout the study, up to 24 months.
  Score change of WHOQOL-BREF from baseline.

CONTACTS AND LOCATIONS:
Locations (1):
- Institute for Clinical and Experimental Medicine, Prague, Czechia